CLINICAL TRIAL: NCT02449928
Title: Peking Union Medical College Hospital, Peking Union Medical College, Chinese Academy of Medical Sciences,
Brief Title: Using Sodium Lactate Ringer's Injection Resuscitate Septic Shock Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PekingUMCH
Record Dates: First submitted 2015-05-18; First posted 2015-05-20 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Severe Sepsis With Septic Shock; Lactate
Keywords: Severe Sepsis with Septic Shock, Lactate

ARMS (2):
- lactate group, (Active Comparator)
  Interventions: Drug: sodium lactate Ringer's injection(Baxter, ShangHai, China)
- control group (Active Comparator)
  Interventions: Drug: Compound Sodium Chloride Injection (CR Double-Crane, Beijing, China)

INTERVENTIONS:
Drug: sodium lactate Ringer's injection(Baxter, ShangHai, China) — use sodium lactate Ringer's injection to resuscitate the septic shock patients(lactate group)
  Arms: lactate group,
Drug: Compound Sodium Chloride Injection (CR Double-Crane, Beijing, China) — use Compound Sodium Chloride injection to resuscitate the septic shock patients(control group)
  Arms: control group

SUMMARY:
Using sodium lactate Ringer's injection resuscitate septic shock patients and Compared with other solution, in order to make clear whether can improve the prognosis.

DETAILED DESCRIPTION:
Experimental evidence repeatedly demonstrated that the shock patients can use substrates other than glucose to sustain increased activity, including lactate.Increased lactate can be the consequence of anaerobic metabolism, i.e., the formation of lactate in the presence of low oxygen. However, emerging evidence demonstrated that in patients with sepsis increased lactate seems predominantly non-hypoxic/ischemic and rather the consequence of increased glycolysis. Utilization of lactate as an alternative fuel may be an adaptive response to maximize energy function and limit substrate reduction.Uptake of exogenous lactate has indeed been demonstrated after traumatic brain injury and acute heart failure in humans.

The investigators assume that administration of supplemental lactate significantly contributes to energy metabolism in septic shock, which can have beneficial help for septic shock resuscitation.

Inclusion criteria:diagnosis in patients with septic shock and age 18 years old or more. Exclusion criteria: pregnant women and nursing mothers, severe liver failure with child class C , use linezolid anti-infection treatment, pheochromocytoma patients, CVVH therapy patients, malignant tumor patients, using epinephrine.

The investigators will use sodium lactate Ringer's injection resuscitate septic shock patients and Compared with other solution, the organ function monitoring include heart, kidney,and brain. Others study endpoints include 28-day mortality,hospitalized mortality.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis in patients with septic shock

Exclusion Criteria:

* pregnant women and nursing mothers
* severe liver failure with child class C
* using Linezolid
* pheochromocytoma
* hematologic malignancy
* using epinephrine
* during CVVH treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2015-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28 days after the diagnosis of septic shock

CONTACTS AND LOCATIONS:
Overall Officials: Da-Wei Liu, Professor, Study Chair — Department of Critical Care Medicine, Peking Union Medical College Hospital